CLINICAL TRIAL: NCT04772235
Title: Phase I Clinical Study to Assess Safety and Efficacy of Repotrectinib Combined With Osimertinib in Patients With Advanced, Metastatic EGFR Mutant NSCLC (TOTEM).
Brief Title: Phase I Study of Repotrectinib and Osimertinib in NSCLC Patients
Acronym: TOTEM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto Oncológico Dr Rosell (Other)
Collaborators: Turning Point Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IOR-TPT-IST-002; 2020-005151-20 (EudraCT Number)
Record Dates: First submitted 2021-02-17; First posted 2021-02-26 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Nsclc
Keywords: Advanced and/or metastatic; EGFR mutant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — repotrectinib; osimertinib

STUDY DESIGN:
Intervention Model Description: This is a single arm, open-label, non-randomized Phase I study with a first dose escalation phase in 3 cohorts to find the RP2D and MTD followed by an expansion phase at the RP2D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced and/or metastatic EGFR mutant NSCLC (Experimental): Eligible advanced and/or metastatic EGFR mutant NSCLC patients will receive the combination of osimertinib and repotrectinib.
  Interventions: Drug: Repotrectinib; Drug: Osimertinib

INTERVENTIONS:
Drug: Repotrectinib — Repotrectinib will be taken orally once daily with or without food Part A: Dose escalation phase, with 3 dose levels for repotrectinib: (1) 80 mg QD, (2) 160 mg QD and (3) 160 mg QD for 14 days followed by 160 mg BID; in combination with 80 mg QD of osimertinib
  Part B: at the RP2D for all patients in combination with osimertinib.
  Other Names: TPX-0005
Drug: Osimertinib — Osimertinib will be taken orally at 80 mg once daily with or without food. Part A: lead in dose in monotherapy at 80 mg QD during 14 days. In combination with repotrectinib afterwards. Depending on the safety and PK/ dose dependent interactions (DDIs) readout during the DLT assessment period, osimertinib dose may be adjusted.
  Part B: at the RP2D level in combination with repotrectinib
  Other Names: Tagrisso

SUMMARY:
This is a Phase I study of repotrectinib in combination with osimertinib in patients with advanced or metastatic EGFR mutant non small cell lung cancer (NSCLC).

The study will be conducted in 2 parts, Part Ia and Part Ib, and its purpose will be to find the incidence of dose-limiting toxicities (DLTs) as defined by the primary safety and tolerability endpoint. The Phase Ia study will also determine the impact of repotrectinib on osimertinib pharmacokinetics (PK) and the maximum tolerated dose (MTD), if reached, of repotrectinib given in combination with osimertinib and the recommended Phase II dose (RP2D). Dose escalation will be conducted according to a 'Rolling-6' based study design with 3 dose levels for repotrectinib: 80 mg once a day (QD), 160 mg QD or 160 mf QD during 14 days followed by 160 mg twice a day (BID); in combination with 80 mg QD of osimertinib. A total of 6 patients will be enrolled in each dose level cohort.

In addition, this Phase Ib study will test early drug activity (efficacy) of the proposed combination treatment in an expansion cohort at the RP2D.

DETAILED DESCRIPTION:
Osimertinib is a third-generation epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI) designed to inhibit activating EGFR mutations (exon 19 deletion and L858R) and resistant T790M mutations with low activity against wild type EGFR. Repotrectinib, potently inhibits Anaplastic Lymphoma Kinase (ALK), Ros proto-oncogene 1 (ROS1), and Tropomyosin receptor kinases (TRK) family kinases; this novel target drug also inhibits Janus kinase 2 (JAK2), sarcoma (SRC), and focal adhesion (FAK), which have shown to be important targets associated with EGFR TKI resistance.

This is a Phase I study of repotrectinib in combination with osimertinib in patients with advanced or metastatic EGFR mutant NSCLC. The study will be conducted in 2 parts, Part Ia and Part Ib:

Part A: of the Phase I study will enroll approximately 9-18 patients in up to 3 dose levels of 3-6 patients each: 80 mg once a day (QD), 160 mg QD or 160 mf QD during 14 days followed by 160 mg twice a day (BID); in combination with 80 mg QD of osimertinib. Patients will receive the combination treatment daily in 3-week cycles until disease progression occurs.

Part B: of the Phase I study is a dose expansion to assess additional PK and safety parameters. Part B will enroll between 20 and 30 patients in 2 cohorts of at least 10 patients each. The 2 cohorts are defined by treatment history: Cohort I, those who have progressed on osimertinib; Cohort II, those who progressed on any first or second generation TKI.

The phase 1A portion of this study will test the safety, tolerability, PK effects, and preliminary efficacy of the EGFR TKI inhibitor osimertinib in combination with repotrectinib in adult patients with advanced/metastatic EGFR mutant NSCLC. The phase 1B (expansion cohort) of this study will test the efficacy of the combination of osimertinib and repotrectinib in terms of progression-free survival and response rate in EGFR TKI-naïve patients with EGFR mutant NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age ≥18.
2. Histological or cytological confirmation of locally advanced or metastatic, non-squamous cell lung carcinoma (NSCLC) in patients who are not candidates for local curative treatment through radical surgery and/or radiotherapy.
3. Stage IV, according to Tumor-nodes-metastasis (TNM) Version 8, including M1a (malignant effusion) or M1b (distant metastasis), or locally advanced disease for which there is no curative treatment (including patients who progress after chemoradiotherapy in Stage III disease).
4. Patients must have been locally diagnosed with EGFR activating mutation (including exon 18, exon 19, exon 21 and mutation T790M) based on FDA approved test (or a local equivalent laboratory developed) test (LDT)). Confirmatory central review will be performed for all patients, in case of discrepancy on EGFR status, central review will prevail.
5. Eastern cooperative oncology group (ECOG) performance status 0-1.
6. Existence of measurable or evaluable disease (according to RECIST 1.1 criteria).
7. Patients with asymptomatic central nervous system (CNS) metastases (treated or untreated) and/or asymptomatic leptomeningeal carcinomatosis are eligible to enroll if they satisfy the following criteria:

   * Patients requiring steroids at a stable or decreasing dose (≤ 12 mg/day dexamethasone or equivalent) for at least 14 days are eligible. Patients on stable doses of levetiracetam (same dose for 14 days) are eligible to be enrolled.
   * A minimum of 14 days must have elapsed from the completion of whole brain radiation treatment (WBRT) before the start of treatment with repotrectinib, and all side effects (with the exception of alopecia) from WBRT are resolved to CTCAE grade ≤ 1.
8. Having available tumor tissue samples, via a biopsy or surgical resection of the primary tumor or metastatic tumor tissue, within 60 days prior to the start of treatment.
9. Life expectancy ≥12 weeks, as determined by a physician.
10. Adequate hematological function, defined as: absolute neutrophil count (ANC) >1.5 x 109/L, platelet count >100.0 x 109/L, and hemoglobin >9.0 g/dL (transfusion allowed at baseline).
11. Adequate liver function, defined as: total bilirubin <1.5 x upper limit of normal (ULN), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) <2.5 x ULN.
12. Adequate renal function, defined as: calculated (Cockcroft-Gault formula) or measured creatinine clearance >50 mL/min and proteinuria <2+ (dipstick).
13. Ability to take part in all study procedures, per investigators.
14. Prior cytotoxic chemotherapy and prior immunotherapy (e.g., anti-PD-1, anti-programmed death ligand 1 (PDL1), anti-T cell immunoglobulin and mucin domain- containing protein 3 (TIM3), anti-OX40) for advanced or metastatic disease is allowed if:

    * At the time of starting treatment with repotrectinib, at least 14 days or 5 half-lives (whichever is shorter) must have elapsed after discontinuation of prior therapy (or at least 42 days for prior nitrosoureas, mitomycin C, and liposomal doxorubicin).
    * All side effects from prior treatments must have resolved to grade ≤ 1 (NCI CTCAE Version 5.0) with the exception of alopecia or other side effects that the investigator does not consider to be a risk to patient safety.
    * Patients with advanced solid tumors harboring ALK, ROS1, neurotrophic tyrosine kinase (NTRK) 1, 2, or 3 rearrangements are eligible if at the time of starting treatment at least 14 days or 5 half-lives (whichever is shorter) have elapsed after discontinuation of prior therapy.
    * There is no limit to the number of prior chemotherapies, immunotherapy, or TKI regimens.
15. All women of childbearing potential (WOCBP), must agree to use highly effective contraception methods during the study treatment period and for at least 2 months after the last dose of EGFR TKI. Male partners of female (WOCBP) patients agree to use condoms during the study and for 2 months after the last dose. Male patients with female partners of WOCBP should use condom protection for 6 months in addition to their female partner (WOCBP) using highly effective contraceptive methods for 4 months after the last dose. Sexually active men, and women of childbearing potential, who are unwilling to use a contraception method are not eligible for the study.
16. Provision of written informed consent, signed and dated by the patient and the investigator, before any study interventions are performed.
17. Part B expansion cohorts only (after the RP2D has been identified):

    * Disease progression following osimertinib with no evidence of tertiary EGFR mutation (i.e., C797S) or MET amplification.
    * Disease progression following first or second generation EGFR TKI (for example, erlotinib,gefitinib, afatinib, dacomitinib) regardless of T790M status.

Exclusion Criteria:

1. Prior exposure to repotrectinib.
2. Diagnosis with any other lung cancer subtype apart from adenocarcinoma including patients with mixed NSCLC with predominantly squamous cell cancer, or with any small-cell lung cancer component, or a tertiary mutation.
3. Presence or history of any other primary malignancy other than NSCLC within 5 years prior to enrollment into the study.
4. Patients with a history of adequately treated basal or squamous cell carcinoma of the skin or any adequately treated in situ carcinoma may be included in the study.
5. Presence of only one measurable or evaluable tumor lesion that has already been resected or irradiated prior to enrollment in the study.
6. Known presence of EGFR exon 20 insertion mutation based on most recent applicable molecular testing.
7. Clinically significant cardiovascular disease (either active or within 6 months prior to enrollment): myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association Classification Class ≥ II), cerebrovascular accident or transient ischemic attack, symptomatic bradycardia, requirement for anti-arrhythmic medication. Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2.
8. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (ECG interval measured from the onset of the QRS complex to the end of the T wave) for heart rate (QTc) > 470 msec obtained from 3 ECGs, using the screening clinic ECG machine-derived QTc value
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval > 250 msec)
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or any concomitant medication known to prolong the QT interval
9. Known active infections requiring ongoing treatment (bacterial, fungal, viral including HIV positivity).
10. Gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would impact on drug absorption.
11. Peripheral neuropathy ≥ grade 2.
12. History of extensive, disseminated, bilateral, or presence of CTCAE grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis. Patients with a history of prior radiation pneumonitis are not excluded.
13. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study or could compromise the protocol objectives in the opinion of the Investigator.
14. For Part B expansion cohorts only (after the RP2D has been identified), presence of a tertiary EGFR mutation (i.e., GFR C797S) mutations and hepatocyte growth factor receptor (MET) amplification.
15. Current use or anticipated need for drugs that are known to be strong Cytochrome P450, family 3, subfamily A (CYP3A) inhibitors or inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Throughout the study period. Approximately 48 months
  Number of patients experiencing AEs, both non treatment related and treatment related, classified by severity and graded according to the NCI CTCAE v5.0
Incidence of Dose limiting toxicities (DLTs) | During the treatment cycle 1, 21 days
  Number of patients experiencing AEs that have been predefined as DLTs: Toxicities resulting in an excessive number of missed doses, Hematologic, renal, hepatic toxicities grade ≥ 3; during the DLT observation period (Cycle 1, 21 days). Only patients in the Part A (dose escalation) of the study.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Throughout the study period. Approximately 48 months
  The ORR will be defined as the proportion of patients with complete response (CR) or partial response (PR). A confirmed response is a response that persists on a repeat-imaging performed at least 4 weeks after initial documentation of the response. Patients with a confirmed objective response (CR or PR) will be referred to as responders. Non-responders will include patients without a confirmed objective response, stable disease (SD), not evaluable (NE), or progression disease (PD). Blinded independent central review (BICR)-confirmed ORR will serve as the secondary (optional) analysis.
Complete response rate (CR) | Throughout the study period. Approximately 48 months
  Number of patients that achieve a confirmed complete response according to RECIST 1.1 criteria. (PR). A confirmed response is a response that persists on a repeat-imaging performed at least 4 weeks after initial documentation of the response.
Partial response rate (PR) | Throughout the study period. Approximately 48 months
  Number of patients that achieve a confirmed partial response according to RECIST 1.1 criteria. (PR). A confirmed response is a response that persists on a repeat-imaging performed at least 4 weeks after initial documentation of the response.
Clinical Benefit Rate (CBR) | Throughout the study period. Approximately 48 months
  The CBR will be defined as the proportion of patients with CR, PR, or stable disease. Stable disease refers to a condition where the tumor is neither increasing nor decreasing in extent or severity for at least 6 weeks after the first dose of repotrectinib, per RECIST, v1.1. The CBR and its 95% CI will be estimated using Clopper-Pearson exact confidence interval (CI).
Duration of Response (DoR) | Throughout the study period. Approximately 48 months
  The DOR will be defined from the first date of objective response (either CR or PR) to the first documentation of radiographically-confirmed disease progression, per RECIST v1.1 guideline and will be censored by the last tumor assessment date for patients without radiologically-confirmed disease progression. The DOR will be calculated only for patients with a confirmed, objective tumor response (PR or CR).
Progression free survival (PFS) | Throughout the study period. Approximately 48 months
  Progression-free survival (PFS) will be defined as the time from the first dose of repotrectinib to the first radiographically-confirmed case of disease progression or to death due to any cause, whichever occurs first. Investigator assessment will serve as the primary efficacy for radiographically-confirmed PFS. BICR-confirmed PFS will serve as the secondary (optional) analysis
Overall survival (OS) | Throughout the study period. Approximately 48 months
  Overall survival (OS) will be defined as the time from first dose of repotrectinib to the date of death, or lost to follow up, whichever occurs first.
Intracranial Objective Response Rate (IC-ORR) | Throughout the study period. Approximately 48 months
  IC-ORR is defined as the proportion of patients with intracranial target lesions that are measurable at Baseline who achieve a PR or CR, per RECIST, v.1.1.
Maximum plasma concentration (Cmax) | on 6 occasions for each patient throughout study: cycle 1 day -1, cycle 1 day 1, cycle 1 day 8, cycle 1 day 15, cycle 2 day 1 and cycle 5 day 1
  Pharmacokinetics (PK) parameter of osimertinib and repotrectinib. Cmax is the maximum (or peak) serum concentration that the drug achieves in blood after the drug has been administered.
Tmax | on 6 occasions for each patient throughout study: cycle 1 day -1, cycle 1 day 1, cycle 1 day 8, cycle 1 day 15, cycle 2 day 1 and cycle 5 day 1
  Pharmacokinetics (PK) parameter of osimertinib and repotrectinib. Tmax is defined as the time of maximum concentration of the drug in blood observed after a drug dose administration.
Area under the curve (AUC) | on 6 occasions for each patient throughout study: cycle 1 day -1, cycle 1 day 1, cycle 1 day 8, cycle 1 day 15, cycle 2 day 1 and cycle 5 day 1
  Pharmacokinetics (PK) parameter of osimertinib and repotrectinib. AUC is the definite integral of a curve that describes the variation of a drug concentration in blood plasma as a function of time. AUC reflects the actual body exposure to drug after administration of a dose.

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Aguilar Hernández, M.D., Study Chair — Institute of oncology Dr. Rosell
Locations (4):
- Spain (4):
  - Hospital Regional Universitario de Málaga, Málaga, Andalusia
  - Hospital Son Espases, Palma, Balearic Islands
  - Quiron Dexeus, Barcelona, Catalonia
  - Hospital Universitario Gregorio Marañón, Madrid

IPD SHARING:
Plan to Share IPD: No